CLINICAL TRIAL: NCT04422093
Title: OrthoKontrol - System Zur Überwachung Der Tragedauer Von kieferorthopädischen Gummizügen
Brief Title: Monitoring System for the Wearing of Orthodontic Elastics
Acronym: OK
Status: Withdrawn | Type: Observational
Why Stopped: The device was found to be too bulky, and therefore we decided not to enrol any subjects.
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: OrthoKontrol
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Medical Device Complication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: OrthoKontrol — Fixing OrthoKontrol Sensor on multibracket appliance to measure cooperation

SUMMARY:
The aim of the study is to validate a novel sensor intended to measure the wearing time of orthodontic elastics in patients with multibracket appliances. The newly developped sensor will be tested in 42 patients over a period of 6 months

DETAILED DESCRIPTION:
Fixed multibracket appliances are used to correct tooth and jaw malocclusions. Usually, elastics are inserted between the upper and lower jaws to adjust the position of the jaws in relation to each other. The wearing time of the elastics determines the duration of the treatment and the quality of the treatment results. While micro-sensors are increasingly used for removable appliances to monitor patient compliance, there is still no such possibility for fixed appliances. This gap is to be closed with the planned 'OrthoKontrol' (intraoral mini-sensor). This is intended to measure and record the wearing time of the elastics.

ELIGIBILITY:
Inclusion Criteria:

* Multibracket appliances (fixed braces) in both jaws
* Need for intermaxillary elastics on at least one side
* Minimum motor skills

Exclusion Criteria:

* Patients with general diseases
* Patients with inflammatory oral diseases
* Patients with physical disabilities, which make it impossible to cooperate
* Independent insertion of the elastics is not possible
* Patients with impaired judgment Pregnant women

Min Age: 11 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with class II malocclusion in treatment with fixed appliances
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
comfort of the device | 6 months
  The wearing comfort for the patient is ok/not ok
Handling of the device | 6 months
  The handling for the therapist is ok/not ok

SECONDARY OUTCOMES:
cooperation | 6 months
  read on the sensors how long the patients followed the instructions

CONTACTS AND LOCATIONS:
Overall Officials: Carlalberta Verna, Principal Investigator — University Center for Dental Medicine, Basel, Switzerland
Locations (1):
- University Center for Dental Medicine UZB, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Mizrahi E. Risk management in clinical practice. Part 7. Dento-legal aspects of orthodontic practice. Br Dent J. 2010 Oct 23;209(8):381-90. doi: 10.1038/sj.bdj.2010.926. PMID 20966997
- [Background] Al-Moghrabi D, Salazar FC, Pandis N, Fleming PS. Compliance with removable orthodontic appliances and adjuncts: A systematic review and meta-analysis. Am J Orthod Dentofacial Orthop. 2017 Jul;152(1):17-32. doi: 10.1016/j.ajodo.2017.03.019. PMID 28651764
- [Background] Huanca Ghislanzoni L, Ameur S, Antonarakis GS, Kiliaridis S. Headgear compliance as assessed by a temperature-sensitive recording device: a prospective clinical study. Eur J Orthod. 2019 Nov 15;41(6):641-645. doi: 10.1093/ejo/cjz036. PMID 31143922
- [Background] Schott TC, Goz G. Applicative characteristics of new microelectronic sensors Smart Retainer(R) and TheraMon(R) for measuring wear time. J Orofac Orthop. 2010 Sep;71(5):339-47. doi: 10.1007/s00056-010-1019-3. Epub 2010 Oct 21. English, German. PMID 20963543